CLINICAL TRIAL: NCT01590810
Title: A Single Rising Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8150
Brief Title: A Single Rising Dose Study of MK-8150 (MK-8150-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8150-001; 2012-001281-15 (EudraCT Number)
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Isolated Systolic Hypertension (ISH)
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension | interventions — MK-8150

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel A-Healthy (Experimental): Within each of the 5 treatment periods, 6 participants will be randomly assigned to receive MK-8150, and 2 will be randomly assigned to receive matching placebo according to a computer-generated allocation schedule. The dose range of MK-8150 for Panel A will be 2.0 mg to 90 mg.
  Interventions: Drug: MK-8150 2.0 mg; Drug: MK-8150 10 mg; Drug: MK-8150 40 mg; Drug: MK-8150 90 mg; Drug: Placebo for MK-8150
- Panel B-Healthy (Experimental): Within each of the 5 treatment periods, 6 participants will be randomly assigned to receive MK-8150, and 2 will be randomly assigned to receive matching placebo according to a computer-generated allocation schedule. The dose range of MK-8150 for Panel B will be 5.0 mg to 160 mg.
  Interventions: Drug: MK-8150 5.0 mg; Drug: MK-8150 20 mg; Drug: MK-8150 60 mg; Drug: MK-8150 120 mg; Drug: MK-8150 160 mg; Drug: Placebo for MK-8150
- Panel C-Mild/Moderate Hypertension (Experimental): Within each of the 5 treatment periods, 6 participants will be randomly assigned to receive MK-8150, and 2 will be randomly assigned to receive matching placebo according to a computer-generated allocation schedule. The dose range of MK-8150 for Panel C will be 160 mg to 1200 mg.
  Interventions: Drug: MK-8150 160 mg; Drug: MK-8150 320 mg; Drug: MK-8150 600 mg; Drug: MK-8150 900 mg; Drug: MK-8150 1200 mg; Drug: Placebo for MK-8150
- Panel D-Healthy (Experimental): Within each panel, 8 subjects will be randomly assigned to MK-8150 and 2 subjects will be randomly assigned to placebo throughout the 5 periods according to a computer-generated allocation schedule. The dose range of MK-8150 for Panel D will be 50 mg to 500 mg.
  Interventions: Drug: Placebo for MK-8150; Drug: MK-8150 50 mg; Drug: MK-8150 100 mg; Drug: MK-8150 200 mg; Drug: MK-8150 400 mg; Drug: MK-8150 500 mg

INTERVENTIONS:
Drug: MK-8150 2.0 mg — Single oral 2.0-mg dose of MK-8150
  Arms: Panel A-Healthy
Drug: MK-8150 10 mg — Single oral 10-mg dose of MK-8150
  Arms: Panel A-Healthy
Drug: MK-8150 40 mg — Single oral 40-mg dose of MK-8150 without food (fasted) and with food (fed)
  Arms: Panel A-Healthy
Drug: MK-8150 90 mg — Single oral 90-mg dose of MK-8150
  Arms: Panel A-Healthy
Drug: MK-8150 5.0 mg — Single oral 5.0-mg dose of MK-8150
  Arms: Panel B-Healthy
Drug: MK-8150 20 mg — Single oral 20-mg dose of MK-8150
  Arms: Panel B-Healthy
Drug: MK-8150 60 mg — Single oral 60-mg dose of MK-8150
  Arms: Panel B-Healthy
Drug: MK-8150 120 mg — Single oral 120-mg dose of MK-8150
  Arms: Panel B-Healthy
Drug: MK-8150 160 mg — Single oral 160-mg dose of MK-8150
  Arms: Panel B-Healthy; Panel C-Mild/Moderate Hypertension
Drug: MK-8150 320 mg — Single oral 320-mg dose of MK-8150
  Arms: Panel C-Mild/Moderate Hypertension
Drug: MK-8150 600 mg — Single oral 600-mg dose of MK-8150
  Arms: Panel C-Mild/Moderate Hypertension
Drug: MK-8150 900 mg — Single oral 900-mg dose of MK-8150
  Arms: Panel C-Mild/Moderate Hypertension
Drug: MK-8150 1200 mg — Single oral 1200-mg dose of MK-8150
  Arms: Panel C-Mild/Moderate Hypertension
Drug: Placebo for MK-8150 — Single oral dose-matched dose of Placebo for MK-8150
Drug: MK-8150 50 mg — Single oral 50-mg dose of MK-8150
  Arms: Panel D-Healthy
Drug: MK-8150 100 mg — Single oral 100-mg dose of MK-8150
  Arms: Panel D-Healthy
Drug: MK-8150 200 mg — Single oral 200-mg dose of MK-8150
  Arms: Panel D-Healthy
Drug: MK-8150 400 mg — Single oral 400-mg dose of MK-8150
  Arms: Panel D-Healthy
Drug: MK-8150 500 mg — Single oral 500-mg dose of MK-8150
  Arms: Panel D-Healthy

SUMMARY:
This study will evaluate the safety and tolerability of MK-8150 and its effect on central systolic blood pressure (cSBP) and heart rate corrected augmentation index (AIx) when given as single oral doses in healthy males and in males with mild-to-moderate hypertension. A primary study hypothesis is that post dose mean change from baseline of time-weighted average across 24 hours (TWA0-24hrs) cSBP or AIx is reduced in participants administered MK-8150 compared to placebo in males with mild to moderate hypertension. A mean decrease from baseline compared to placebo of ≥5 mm Hg in TWA0-24hrs cSBP or of ≥5 percentage points in TWA0-24hrs AIx is considered clinically meaningful.

DETAILED DESCRIPTION:
Up to three planned panels (A, B and C) of either 8 healthy participants or 8 participants with mild to moderate hypertension will be enrolled. For Panel A and Panel B, dosing will occur in an alternating fashion between Panel A and Panel B with dosing commencing in Panel A. Participants will receive alternating single rising oral doses of MK-8150 or placebo in up to 5 treatment periods (Periods 1 through 5). Subsequent doses in any Panel will be administered only after careful evaluation of safety, tolerability, and pharmacodynamic effects of a given dose. For Panel C, participants will receive single rising oral doses of MK-8150 or placebo in up to 5 treatment periods (Periods 1 through 5). Depending on safety, tolerability and hemodynamic effects observed in the healthy participants, Panels A and/or B may be truncated and dosing may proceed in Panel C with hypertensive participants. In this case, dosing of hypertensive participants in Panel C will start with the second highest dose achieved in healthy participants.

Amendment 1 of the protocol added Panel D (healthy males) based on the pharmacokinetic, pharmacodynamic and safety results from Panels A-C. Participants in Panel D will receive single rising oral doses of MK-8150 or placebo in up to 5 treatment periods (Periods 1 through 5) at a dose range of 50 mg to 500 mg of MK-8150. Each treatment period will be approximately 3-4 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age for Panels A, B and D, or between 18 and 60 years of age (inclusive) for Panel C.
* Systolic blood pressure (SBP) > 110 and ≤ 140 mmHg for Panels A, B, and D or SBP values of 140-175 mmHg and diastolic blood pressure (DBP) of 90-105 mmHg on at least three different occasions at the prestudy (screening) visit for Panel C. Participants being treated with medication for their hypertension may be included as long as they are titrated off of their medication
* Body Mass Index (BMI) ≥ 18 kg/m^2 and ≤ 32 kg/m^2
* Healthy (with the exception of hypertensive subjects in Panel C)
* No clinically significant abnormality on electrocardiogram (ECG)
* No history of clinically significant cardiac disease
* No history of heart failure
* Nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion Criteria:

* Mentally or legally incapacitated
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular (except mild to moderate hypertension), hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Functional disability that can interfere with rising from a sitting position to the standing position
* History of neoplastic disease (cancer)
* Unable to refrain from or anticipates the use of any medication during the study
* Anticipates using medication for erectile dysfunction during the study
* Uses or anticipates using organic nitrates during the study (e.g. nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, pentaerythritol)
* Anticipates using cytochrome P450 inhibitors (e.g. ketoconazole) or inducers (e.g. rifampin) during the study
* Consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, or other caffeinated beverages per day
* Has had major surgery, donated or lost 1 unit of blood or participated in another investigational study within 4 weeks
* History of significant multiple and/or severe allergies (including latex allergy)
* Regular user (including recreational user) of illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05-07 (Actual); Primary Completion 2013-01-24 (Actual); Study Completion 2013-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Knox CD, de Kam PJ, Azer K, Wong P, Ederveen AG, Shevell D, Morabito C, Meehan AG, Liu W, Reynders T, Denef JF, Mitselos A, Jonathan D, Gutstein DE, Mitra K, Sun SY, Lo MM, Cully D, Ali A. Discovery and Clinical Evaluation of MK-8150, A Novel Nitric Oxide Donor With a Unique Mechanism of Nitric Oxide Release. J Am Heart Assoc. 2016 Aug 25;5(9):e003493. doi: 10.1161/JAHA.116.003493. PMID 27561272
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8150-001&kw=8150-001&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A - MK-8150 2 to 90 mg/Placebo: Within each of the up to 5 treatment periods in Panel A, 6 healthy participants were randomly assigned to receive a single dose of MK-8150, and 2 were randomly assigned to receive single administration of matching placebo according to a computer-generated allocation schedule. By protocol allocation schedule participants did not have fixed assignment to single dose MK-8150 or placebo for all treatment periods, but were reallocated from one treatment period to the next, so that a participant could receive both MK-8150 and placebo, in different periods of the Panel. The dose range of MK-8150 administered for Panel A was 2 mg to 90 mg.
- Panel B - MK-8150 4 to 120 mg/Placebo: Within each of the up to 5 treatment periods in Panel B, 6 healthy participants were randomly assigned to receive a single dose of MK-8150, and 2 were randomly assigned to receive single administration of matching placebo according to a computer-generated allocation schedule. By protocol allocation schedule participants did not have fixed assignment to single dose MK-8150 or placebo for all treatment periods, but were reallocated from one treatment period to the next, so that a participant could receive both MK-8150 and placebo, in different periods of the Panel. The dose range of MK-8150 administered for Panel B was 4 mg to 120 mg.
- Panel C - MK-8150 5 to 90 mg/Placebo: Within each of the up to 5 treatment periods in Panel C, 6 participants with mild to moderate hypertension were randomly assigned to receive a single dose of MK-8150, and 2 were randomly assigned to receive single administration of matching placebo according to a computer-generated allocation schedule. By protocol allocation schedule participants did not have fixed assignment to single dose MK-8150 or placebo for all treatment periods, but were reallocated from one treatment period to the next, so that a participant could receive both MK-8150 and placebo, in different periods of the Panel. The dose range of MK-8150 administered for Panel C was 5 mg to 90 mg.
- Panel D - MK-8150 50 to 200 mg: Description: Within Panel D, 8 healthy participants were randomly assigned to receive single doses of MK-8150, and 2 were randomly assigned to receive single administrations of matching placebo throughout the up to 5 treatment periods according to a computer-generated allocation schedule (i.e., assignment of a participant to either MK-8150 or placebo was fixed for all Panel D periods). This reporting group presents data for the Panel D participants administered MK-8150. The dose range of MK-8150 administered for Panel D was 50 mg to 200 mg.
- Panel D - Placebo: Within Panel D, 8 healthy participants were randomly assigned to receive single doses of MK-8150, and 2 were randomly assigned to receive single administrations of matching placebo throughout the up to 5 treatment periods according to a computer-generated allocation schedule (i.e., assignment of a participant to either MK-8150 or placebo was fixed for all Panel D periods). This reporting group presents data for the Panel D participants administered placebo.
Period: Overall Study
Arm/Group | Panel A - MK-8150 2 to 90 mg/Placebo | Panel B - MK-8150 4 to 120 mg/Placebo | Panel C - MK-8150 5 to 90 mg/Placebo | Panel D - MK-8150 50 to 200 mg | Panel D - Placebo
Started | 8 | 8 | 8 | 8 | 2
Completed | 8 | 7 | 7 | 8 | 2
Not Completed | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A - MK-8150 2 to 90 mg/Placebo | Panel B - MK-8150 4 to 120 mg/Placebo | Panel C - MK-8150 5 to 90 mg/Placebo | Panel D - MK-8150 50 to 200 mg | Panel D - Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (9.8) | 34.8 (8.0) | 51.4 (6.8) | 44.1 (6.9) | 39.0 (12.7) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 2 | 34
Central Systolic Blood Pressure (cSBP) [Mean (Standard Deviation); unit: mm Hg] | 98 (7) | 98 (6) | 125 (8) | 102 (9) | 105 (6) | 106 (13)
Augmentation Index (AIx) [Mean (Standard Deviation); unit: percentage of central pulse pressure] — AIx was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. AIx is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness.
  percentage of central pulse pressure | 7 (3) | 8 (4) | 22 (8) | 10 (11) | 8 (12) | 12 (9)
Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute] | 58 (7) | 54 (5) | 67 (9) | 61 (7) | 45 (1) | 59 (9)
Central Diastolic Blood Pressure (cDBP) [Mean (Standard Deviation); unit: mm Hg] | 85 (6) | 84 (6) | 107 (6) | 86 (8) | 91 (6) | 91 (11)
Peripheral Systolic Blood Pressure (pSBP) [Mean (Standard Deviation); unit: mm Hg] | 119 (5) | 119 (6) | 148 (7) | 125 (8) | 126 (12) | 128 (14)
Peripheral Diastolic Blood Pressure (pDBP) [Mean (Standard Deviation); unit: mm Hg] | 75 (6) | 73 (6) | 94 (6) | 75 (8) | 80 (7) | 79 (10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study drug, is also an AE.
Time Frame: Up to 14 days after the last dose (Up to approximately 42 days)
Population: All participants who received a dose of study drug
Measure: Number; unit: participants
Arm/Group | Panel A - MK-8150 2 to 90 mg/Placebo | Panel B - MK-8150 4 to 120 mg/Placebo | Panel C - MK-8150 5 to 90 mg/Placebo | Panel D - MK-8150 50 to 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
participants | 8 | 8 | 7 | 7 | 2

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 1
Time Frame: Up to 14 days after the last dose (Up to approximately 42 days)
Population: All participants who received a dose of study drug
Measure: Number; unit: participants
Arm/Group | Panel A - MK-8150 2 to 90 mg/Placebo | Panel B - MK-8150 4 to 120 mg/Placebo | Panel C - MK-8150 5 to 90 mg/Placebo | Panel D - MK-8150 50 to 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Time-weighted Average Across 24 Hours (TWA0-24hrs) cSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: cSBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cSBP value by that cSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population. 2 participants received placebo in period of fasted administration of MK-8150 24 mg dose and again received placebo during the period of fed administration of that dose. Data for both administrations of placebo in these participants are included (i.e., for placebo, analysis includes 10 observations from 8 participants)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel A - MK-8150 2 mg: Single dose of MK-8150 2 mg
- Panel A - MK-8150 6 mg: Single dose of MK-8150 6 mg
- Panel A - MK-8150 24 mg: Single dose of MK-8150 24 mg
- Panel A - MK-8150 24 mg (Fed Condition): Single dose of MK-8150 24 mg, administered following a standard high-fat breakfast (Fed condition). MK-8150 24 mg doses in this Panel A period were the only doses in study administered after a meal. All other doses in study were administered after an overnight fast.
- Panel A - MK-8150 90 mg: Single dose of MK-8150 90 mg
- Panel A - Placebo: Single dose of placebo
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
mm Hg | 1.33 (0.99) | -1.65 (1.31) | -7.69 (1.71) | -6.29 (1.82) | -9.86 (1.66) | 0.55 (1.08)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.503, Mixed Models Analysis; Least Squares (LS) Mean Difference = 0.78, 95% CI 2-sided [-1.59 to 3.15], Standard Error of Mean 1.15 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.20, 95% CI 2-sided [-2.86 to -1.55], Standard Error of Mean 0.32 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.23, 95% CI 2-sided [-10.13 to -6.34], Standard Error of Mean 0.92 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -6.84, 95% CI 2-sided [-9.10 to -4.58], Standard Error of Mean 1.10 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.41, 95% CI 2-sided [-12.89 to -7.92], Standard Error of Mean 1.21 — Difference is MK-8150 dose - placebo

4. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population. 2 participants received placebo in period of initial administration of MK-8150 120 mg dose and again received placebo during the period of repeat administration of that dose. Data for both administrations of placebo in these participants are included (i.e., for placebo, analysis includes 10 observations from 8 participants)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel B - MK-8150 4 mg: Single dose of MK-8150 4 mg
- Panel B - MK-8150 12 mg: Single dose of MK-8150 12 mg
- Panel B - MK-8150 45 mg: Single dose of MK-8150 45 mg
- Panel B - MK-8150 120 mg: Single dose of MK-8150 120 mg
- Panel B - MK-8150 120 mg (Repeat Dose): Single dose of MK-8150 120 mg. This was a repeat administration of the 120 mg dose, permitted under flexible design of protocol
- Panel B - Placebo: Single dose of placebo
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
mm Hg | -5.06 (0.91) | -7.64 (1.50) | -11.67 (1.68) | -14.20 (1.60) | -11.91 (1.26) | -2.18 (1.11)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.052, Mixed Models Analysis; LS Mean Difference = -2.89, 95% CI 2-sided [-5.79 to 0.02], Standard Error of Mean 1.40 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; LS Mean Difference = -5.46, 95% CI 2-sided [-9.49 to -1.43], Standard Error of Mean 1.95 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.49, 95% CI 2-sided [-14.20 to -4.79], Standard Error of Mean 2.27 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.02, 95% CI 2-sided [-16.51 to -7.52], Standard Error of Mean 2.17 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.73, 95% CI 2-sided [-12.93 to -6.53], Standard Error of Mean 1.55 — Difference is MK-8150 dose - placebo

5. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel C - MK-8150 5 mg: Single dose of MK-8150 5 mg
- Panel C - MK-8150 24 mg: Single dose of MK-8150 24 mg
- Panel C - MK-8150 90 mg: Single dose of MK-8150 90 mg
- Panel C - Placebo: Single dose of placebo
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
mm Hg | -11.69 (3.01) | -18.38 (4.47) | -25.11 (3.20) | -7.60 (4.46)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis; LS Mean Difference = -4.10, 95% CI 2-sided [-16.44 to 8.25], Standard Error of Mean 5.61 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis; LS Mean Difference = -10.79, 95% CI 2-sided [-23.37 to 1.79], Standard Error of Mean 5.72 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; LS Mean Difference = -17.51, 95% CI 2-sided [-28.85 to -6.18], Standard Error of Mean 5.15 — Difference is MK-8150 dose - placebo

6. Primary Outcome: Change From Baseline in TWA0-24hrs cSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 3
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population. The same 2 participants received placebo throughout all treatment periods of Panel D. Data for all administrations of placebo in these participants are included (i.e., for placebo, analysis includes 8 observations from 2 participants)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Panel D - MK-8150 50 mg: Single dose of MK-8150 50 mg
- Panel D - MK-8150 50 mg (Repeat Dose): Single dose of MK-8150 50 mg. This was a repeat administration of the 50 mg dose, permitted under flexible design of protocol
- Panel D - MK-8150 100 mg: Single dose of MK-8150 100 mg
- Panel D - MK-8150 200 mg: Single dose of MK-8150 200 mg
- Panel D - Placebo: Single dose of placebo
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
mm Hg | -16.23 (1.40) | -13.22 (1.55) | -15.84 (1.50) | -15.86 (1.47) | -3.02 (0.38)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.21, 95% CI 2-sided [-16.84 to -9.59], Standard Error of Mean 1.74 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.20, 95% CI 2-sided [-13.94 to -6.45], Standard Error of Mean 1.80 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.82, 95% CI 2-sided [-16.45 to -9.19], Standard Error of Mean 1.74 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.84, 95% CI 2-sided [-16.49 to -9.19], Standard Error of Mean 1.75 — Difference is MK-8150 dose - placebo

7. Primary Outcome: Change From Baseline in TWA0-24hrs AIx in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: AIx was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Augmentation index is the percentage of the central pulse pressure attributed to the reflected pulse wave, and is an indirect measure of systemic arterial stiffness. Time-weighted average was obtained as follows: For all AIx values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each AIx value by that AIx value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified AIx value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement. AIx was adjusted for HR.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose; except Period 1: Pre-dose and 2, 4, 12 and 24 hours post dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
percentage of central pulse pressure | -0.75 (1.99) | -0.67 (1.63) | -10.06 (1.62) | -6.59 (2.22) | -15.22 (1.53) | 1.56 (1.32)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis; LS Mean Difference = -2.31, 95% CI 2-sided [-4.73 to 0.11], Standard Error of Mean 1.18 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis; LS Mean Difference = -2.23, 95% CI 2-sided [-4.00 to -0.45], Standard Error of Mean 0.86 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.62, 95% CI 2-sided [-14.42 to -8.82], Standard Error of Mean 1.36 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.15, 95% CI 2-sided [-11.34 to -4.96], Standard Error of Mean 1.55 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -16.78, 95% CI 2-sided [-20.81 to -12.75], Standard Error of Mean 1.96 — Difference is MK-8150 dose - placebo

8. Primary Outcome: Change From Baseline in TWA0-24hrs AIx in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 7
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
percentage of central pulse pressure | -3.04 (1.55) | -6.85 (1.83) | -13.57 (2.54) | -18.42 (1.55) | -16.33 (2.22) | -0.09 (1.50)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; LS Mean Difference = -2.95, 95% CI 2-sided [-5.56 to -0.34], Standard Error of Mean 1.26 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS Mean Difference = -6.76, 95% CI 2-sided [-11.29 to -2.22], Standard Error of Mean 2.19 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.48, 95% CI 2-sided [-20.03 to -6.93], Standard Error of Mean 3.16 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -18.33, 95% CI 2-sided [-21.98 to -14.68], Standard Error of Mean 1.76 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -16.24, 95% CI 2-sided [-20.29 to -12.19], Standard Error of Mean 1.96 — Difference is MK-8150 dose - placebo

9. Primary Outcome: Change From Baseline in TWA0-24hrs AIx in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 7
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
percentage of central pulse pressure | -8.32 (1.69) | -12.09 (3.25) | -21.03 (1.90) | -6.73 (2.49)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.539, Mixed Models Analysis; LS Mean Difference = -1.59, 95% CI 2-sided [-7.12 to 3.93], Standard Error of Mean 2.51 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.113, Mixed Models Analysis; LS Mean Difference = -5.36, 95% CI 2-sided [-12.23 to 1.50], Standard Error of Mean 3.12 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -14.30, 95% CI 2-sided [-19.69 to -8.91], Standard Error of Mean 2.45 — Difference is MK-8150 dose - placebo

10. Primary Outcome: Change From Baseline in TWA0-24hrs AIx in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 7
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage of central pulse pressure
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
percentage of central pulse pressure | -13.83 (1.54) | -12.04 (1.46) | -15.09 (1.12) | -14.42 (1.29) | -1.46 (0.17)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.36, 95% CI 2-sided [-15.62 to -9.11], Standard Error of Mean 1.56 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.58, 95% CI 2-sided [-13.74 to -7.42], Standard Error of Mean 1.51 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.63, 95% CI 2-sided [-16.12 to -11.13], Standard Error of Mean 1.20 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -12.96, 95% CI 2-sided [-15.85 to -10.08], Standard Error of Mean 1.38 — Difference is MK-8150 dose - placebo

11. Primary Outcome: Change From Baseline in Time-weighted Average Across 12 Hours (TWA0-12hrs) HR in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: HR was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all HR values obtained over the 12-hour observation period, multiply the length of time that the participant spent at each HR value by that HR value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified HR value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
beats per minute | 2.94 (1.31) | 4.08 (1.61) | 4.07 (1.47) | 7.54 (2.19) | 4.04 (1.65) | 1.89 (1.43)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; LS Mean Difference = 1.05, 95% CI 2-sided [-0.50 to 2.60], Standard Error of Mean 0.75 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis; LS Mean Difference = 2.18, 95% CI 2-sided [-0.25 to 4.61], Standard Error of Mean 1.18 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = 2.18, 95% CI 2-sided [1.04 to 3.32], Standard Error of Mean 0.55 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 5.64, 95% CI 2-sided [3.14 to 8.15], Standard Error of Mean 1.22 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; LS Mean Difference = 2.15, 95% CI 2-sided [0.63 to 3.67], Standard Error of Mean 0.74 — Difference is MK-8150 dose - placebo

12. Primary Outcome: Change From Baseline in TWA0-12hrs HR in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 11
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
beats per minute | -0.26 (1.10) | -0.91 (1.57) | 0.66 (1.75) | 3.17 (0.91) | 5.19 (1.45) | 0.57 (1.16)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.557, Mixed Models Analysis; LS Mean Difference = -0.83, 95% CI 2-sided [-3.70 to 2.05], Standard Error of Mean 1.39 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.175, Mixed Models Analysis; LS Mean Difference = -1.48, 95% CI 2-sided [-3.65 to 0.70], Standard Error of Mean 1.05 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.951, Mixed Models Analysis; LS Mean Difference = 0.09, 95% CI 2-sided [-3.04 to 3.23], Standard Error of Mean 1.52 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = 2.61, 95% CI 2-sided [1.34 to 3.88], Standard Error of Mean 0.61 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 4.62, 95% CI 2-sided [3.00 to 6.24], Standard Error of Mean 0.78 — Difference is MK-8150 dose - placebo

13. Primary Outcome: Change From Baseline in TWA0-12hrs HR in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 11
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
beats per minute | -6.11 (2.32) | -3.74 (1.58) | -1.02 (1.75) | -4.67 (2.23)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.241, Mixed Models Analysis; LS Mean Difference = -1.45, 95% CI 2-sided [-4.01 to 1.12], Standard Error of Mean 1.16 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.664, Mixed Models Analysis; LS Mean Difference = 0.92, 95% CI 2-sided [-3.63 to 5.48], Standard Error of Mean 2.07 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis; LS Mean Difference = 3.65, 95% CI 2-sided [-1.03 to 8.33], Standard Error of Mean 2.13 — Difference is MK-8150 dose - placebo

14. Primary Outcome: Change From Baseline in TWA0-12hrs HR in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 11
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours post dose
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
beats per minute | -1.24 (1.90) | -1.09 (2.15) | -0.52 (1.59) | 3.83 (2.15) | -5.67 (3.66)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p = 0.385, Mixed Models Analysis; LS Mean Difference = 4.42, 95% CI 2-sided [-5.96 to 14.81], Standard Error of Mean 4.98 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p = 0.385, Mixed Models Analysis; LS Mean Difference = 4.58, 95% CI 2-sided [-6.16 to 15.32], Standard Error of Mean 5.15 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p = 0.276, Mixed Models Analysis; LS Mean Difference = 5.15, 95% CI 2-sided [-4.44 to 14.74], Standard Error of Mean 4.60 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis; LS Mean Difference = 9.50, 95% CI 2-sided [-0.81 to 19.81], Standard Error of Mean 4.94 — Difference is MK-8150 dose - placebo

15. Primary Outcome: Change From Baseline in TWA0-24hrs cDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: cDBP was measured by applanation tonometry of the radial artery, using the SphygmoCor System. The central pressure waveform was determined from the peripheral pressure waveform by a transfer function. Time-weighted average was obtained as follows: For all cDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each cDBP value by that cDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified cDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement.
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
mm Hg | 0.74 (1.07) | -1.97 (1.46) | -8.34 (1.77) | -6.73 (2.27) | -10.54 (1.62) | -0.23 (1.11)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.383, Mixed Models Analysis; LS Mean Difference = 0.97, 95% CI 2-sided [-1.28 to 3.22], Standard Error of Mean 1.09 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS Mean Difference = -1.75, 95% CI 2-sided [-2.79 to -0.70], Standard Error of Mean 0.51 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.11, 95% CI 2-sided [-10.08 to -6.14], Standard Error of Mean 0.96 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.50, 95% CI 2-sided [-9.74 to -3.25], Standard Error of Mean 1.58 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.31, 95% CI 2-sided [-12.84 to -7.78], Standard Error of Mean 1.23 — Difference is MK-8150 dose - placebo

16. Primary Outcome: Change From Baseline in TWA0-24hrs cDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 15
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
mm Hg | -5.02 (1.10) | -7.76 (1.61) | -11.88 (1.75) | -14.12 (1.95) | -12.21 (1.30) | -2.96 (1.33)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.216, Mixed Models Analysis; LS Mean Difference = -2.07, 95% CI 2-sided [-5.43 to 1.30], Standard Error of Mean 1.62 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.046, Mixed Models Analysis; LS Mean Difference = -4.80, 95% CI 2-sided [-9.51 to -0.10], Standard Error of Mean 2.27 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS Mean Difference = -8.93, 95% CI 2-sided [-14.10 to -3.76], Standard Error of Mean 2.50 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -11.16, 95% CI 2-sided [-16.64 to -5.68], Standard Error of Mean 2.65 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.25, 95% CI 2-sided [-12.70 to -5.80], Standard Error of Mean 1.67 — Difference is MK-8150 dose - placebo

17. Primary Outcome: Change From Baseline in TWA0-24hrs cDBP in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 15
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
mm Hg | -10.40 (1.96) | -16.32 (3.97) | -23.65 (2.67) | -8.14 (3.76)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.635, Mixed Models Analysis; LS Mean Difference = -2.27, 95% CI 2-sided [-12.50 to 7.96], Standard Error of Mean 4.65 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.143, Mixed Models Analysis; LS Mean Difference = -8.18, 95% CI 2-sided [-19.58 to 3.22], Standard Error of Mean 5.18 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = -15.51, 95% CI 2-sided [-25.01 to -6.01], Standard Error of Mean 4.32 — Difference is MK-8150 dose - placebo

18. Primary Outcome: Change From Baseline in TWA0-24hrs cDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 15
Time Frame: Pre-dose and 2, 3, 4, 6, 8, 12, 16 and 24 hours post dose
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
mm Hg | -15.55 (1.05) | -13.26 (0.93) | -15.35 (1.19) | -15.84 (1.10) | -4.71 (0.52)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.84, 95% CI 2-sided [-13.79 to -7.89], Standard Error of Mean 1.42 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.55, 95% CI 2-sided [-11.18 to -5.91], Standard Error of Mean 1.26 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.64, 95% CI 2-sided [-13.44 to -7.84], Standard Error of Mean 1.34 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.13, 95% CI 2-sided [-13.97 to -8.29], Standard Error of Mean 1.36 — Difference is MK-8150 dose - placebo

19. Primary Outcome: Change From Baseline in TWA0-24hrs pSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: pSBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pSBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pSBP value by that pSBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pSBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
mm Hg | 0.73 (1.35) | -0.24 (1.45) | -3.13 (1.56) | -1.91 (1.42) | -4.46 (1.70) | 1.46 (1.41)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.547, Mixed Models Analysis; LS Mean Difference = -0.73, 95% CI 2-sided [-3.19 to 1.73], Standard Error of Mean 1.19 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = -1.70, 95% CI 2-sided [-2.79 to -0.62], Standard Error of Mean 0.53 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.59, 95% CI 2-sided [-6.23 to -2.94], Standard Error of Mean 0.80 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -3.37, 95% CI 2-sided [-4.98 to -1.76], Standard Error of Mean 0.78 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -5.92, 95% CI 2-sided [-8.24 to -3.59], Standard Error of Mean 1.13 — Difference is MK-8150 dose - placebo

20. Primary Outcome: Change From Baseline in TWA0-24hrs pSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
mm Hg | -4.61 (1.00) | -6.81 (1.61) | -7.16 (2.00) | -8.50 (1.39) | -6.40 (1.19) | -1.17 (1.01)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis; LS Mean Difference = -3.43, 95% CI 2-sided [-6.19 to -0.67], Standard Error of Mean 1.33 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.64, 95% CI 2-sided [-8.43 to -2.84], Standard Error of Mean 1.35 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS Mean Difference = -5.99, 95% CI 2-sided [-9.94 to -2.04], Standard Error of Mean 1.91 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.33, 95% CI 2-sided [-10.90 to -3.76], Standard Error of Mean 1.73 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -5.22, 95% CI 2-sided [-7.76 to -2.69], Standard Error of Mean 1.22 — Difference is MK-8150 dose - placebo

21. Primary Outcome: Change From Baseline in TWA0-24hrs pSBP in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
mm Hg | -12.32 (3.88) | -18.26 (4.84) | -21.42 (3.63) | -5.39 (6.63)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.311, Mixed Models Analysis; LS Mean Difference = -6.93, 95% CI 2-sided [-21.27 to 7.42], Standard Error of Mean 6.52 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.078, Mixed Models Analysis; LS Mean Difference = -12.87, 95% CI 2-sided [-27.44 to 1.69], Standard Error of Mean 6.62 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis; LS Mean Difference = -16.03, 95% CI 2-sided [-29.87 to -2.19], Standard Error of Mean 6.29 — Difference is MK-8150 dose - placebo

22. Primary Outcome: Change From Baseline in TWA0-24hrs pSBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
mm Hg | -12.77 (1.14) | -10.19 (1.86) | -11.19 (1.78) | -10.47 (1.79) | -3.00 (0.85)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.77, 95% CI 2-sided [-12.90 to -6.65], Standard Error of Mean 1.50 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference = -7.19, 95% CI 2-sided [-11.57 to -2.81], Standard Error of Mean 2.10 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = -8.19, 95% CI 2-sided [-12.40 to -3.98], Standard Error of Mean 2.02 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS Mean Difference = -7.47, 95% CI 2-sided [-11.69 to -3.25], Standard Error of Mean 2.02 — Difference is MK-8150 dose - placebo

23. Primary Outcome: Change From Baseline in TWA0-24hrs pDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel A)
Description: pDBP was measured with a validated automatic measuring device. Time-weighted average was obtained as follows: For all pDBP values obtained over the 24-hour observation period, multiply the length of time that the participant spent at each pDBP value by that pDBP value, add these products together, and then divide by duration of the observation period. The length of time spent at an identified pDBP value was defined as the time elapsed since previous post-dose measurement, or time elapsed since drug administration, if there is no previous post-dose measurement.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel A - MK-8150 2 mg | Panel A - MK-8150 6 mg | Panel A - MK-8150 24 mg | Panel A - MK-8150 24 mg (Fed Condition) | Panel A - MK-8150 90 mg | Panel A - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
mm Hg | -0.92 (0.61) | -2.58 (1.13) | -8.01 (1.56) | -6.69 (2.30) | -9.85 (1.38) | -1.24 (0.90)
Statistical Analysis 1: Comparison: Panel A - MK-8150 2 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.765, Mixed Models Analysis; LS Mean Difference = 0.31, 95% CI 2-sided [-1.82 to 2.45], Standard Error of Mean 1.04 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel A - MK-8150 6 mg vs Panel A - Placebo; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; LS Mean Difference = -1.34, 95% CI 2-sided [-2.49 to -0.20], Standard Error of Mean 0.56 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel A - MK-8150 24 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -6.77, 95% CI 2-sided [-9.18 to -4.36], Standard Error of Mean 1.17 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel A - MK-8150 24 mg (Fed Condition) vs Panel A - Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; LS Mean Difference = -5.45, 95% CI 2-sided [-9.46 to -1.44], Standard Error of Mean 1.95 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel A - MK-8150 90 mg vs Panel A - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.61, 95% CI 2-sided [-11.28 to -5.94], Standard Error of Mean 1.30 — Difference is MK-8150 dose - placebo

24. Primary Outcome: Change From Baseline in TWA0-24hrs pDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel B)
Description: as for outcome 23
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel B - MK-8150 4 mg | Panel B - MK-8150 12 mg | Panel B - MK-8150 45 mg | Panel B - MK-8150 120 mg | Panel B - MK-8150 120 mg (Repeat Dose) | Panel B - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 8
mm Hg | -3.91 (1.02) | -6.21 (1.34) | -9.64 (1.86) | -11.69 (1.85) | -10.20 (1.11) | -1.90 (0.85)
Statistical Analysis 1: Comparison: Panel B - MK-8150 4 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis; LS Mean Difference = -2.02, 95% CI 2-sided [-4.89 to 0.86], Standard Error of Mean 1.39 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel B - MK-8150 12 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis; LS Mean Difference = -4.32, 95% CI 2-sided [-8.40 to -0.24], Standard Error of Mean 1.97 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel B - MK-8150 45 mg vs Panel B - Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; LS Mean Difference = -7.75, 95% CI 2-sided [-12.58 to -2.92], Standard Error of Mean 2.34 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel B - MK-8150 120 mg vs Panel B - Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.79, 95% CI 2-sided [-14.49 to -5.09], Standard Error of Mean 2.27 — Difference is MK-8150 dose - placebo
Statistical Analysis 5: Comparison: Panel B - MK-8150 120 mg (Repeat Dose) vs Panel B - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.31, 95% CI 2-sided [-11.30 to -5.31], Standard Error of Mean 1.45 — Difference is MK-8150 dose - placebo

25. Primary Outcome: Change From Baseline in TWA0-24hrs pDBP in Male Participants With Mild to Moderate Hypertension Administered Single Doses of MK-8150 and Placebo (Panel C)
Description: as for outcome 23
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel C - MK-8150 5 mg | Panel C - MK-8150 24 mg | Panel C - MK-8150 90 mg | Panel C - Placebo
Number analyzed (Participants) | 5 | 5 | 6 | 6
mm Hg | -7.87 (1.89) | -12.90 (3.55) | -19.82 (2.27) | -6.14 (3.80)
Statistical Analysis 1: Comparison: Panel C - MK-8150 5 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.675, Mixed Models Analysis; LS Mean Difference = -1.72, 95% CI 2-sided [-10.54 to 7.09], Standard Error of Mean 4.00 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel C - MK-8150 24 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.174, Mixed Models Analysis; LS Mean Difference = -6.76, 95% CI 2-sided [-16.98 to 3.46], Standard Error of Mean 4.64 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel C - MK-8150 90 mg vs Panel C - Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; LS Mean Difference = -13.68, 95% CI 2-sided [-22.55 to -4.81], Standard Error of Mean 4.03 — Difference is MK-8150 dose - placebo

26. Primary Outcome: Change From Baseline in TWA0-24hrs pDBP in Healthy Male Participants Administered Single Doses of MK-8150 and Placebo (Panel D)
Description: as for outcome 23
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16 and 24 hours post dose
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Panel D - MK-8150 50 mg | Panel D - MK-8150 50 mg (Repeat Dose) | Panel D - MK-8150 100 mg | Panel D - MK-8150 200 mg | Panel D - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 2
mm Hg | -13.91 (0.77) | -11.65 (0.61) | -13.36 (0.87) | -14.31 (0.87) | -4.79 (1.17)
Statistical Analysis 1: Comparison: Panel D - MK-8150 50 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.12, 95% CI 2-sided [-12.22 to -6.03], Standard Error of Mean 1.49 — Difference is MK-8150 dose - placebo
Statistical Analysis 2: Comparison: Panel D - MK-8150 50 mg (Repeat Dose) vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -6.86, 95% CI 2-sided [-9.73 to -3.99], Standard Error of Mean 1.38 — Difference is MK-8150 dose - placebo
Statistical Analysis 3: Comparison: Panel D - MK-8150 100 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.57, 95% CI 2-sided [-11.51 to -5.64], Standard Error of Mean 1.41 — Difference is MK-8150 dose - placebo
Statistical Analysis 4: Comparison: Panel D - MK-8150 200 mg vs Panel D - Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -9.52, 95% CI 2-sided [-12.55 to -6.50], Standard Error of Mean 1.45 — Difference is MK-8150 dose - placebo

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose (Up to approximately 42 days)
Groups:
- Panel D - MK-8150 50 to 200 mg: Within Panel D, 8 healthy participants were randomly assigned to receive single doses of MK-8150, and 2 were randomly assigned to receive single administrations of matching placebo throughout the up to 5 treatment periods according to a computer-generated allocation schedule (i.e., assignment of a participant to either MK-8150 or placebo was fixed for all Panel D periods). This reporting group presents data for the Panel D participants administered MK-8150. The dose range of MK-8150 administered for Panel D was 50 mg to 200 mg.
Arm/Group | Panel A - MK-8150 2 to 90 mg/Placebo | Panel B - MK-8150 4 to 120 mg/Placebo | Panel C - MK-8150 5 to 90 mg/Placebo | Panel D - MK-8150 50 to 200 mg | Panel D - Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 7/8 | 7/8 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A - MK-8150 2 to 90 mg/Placebo (N=8) | Panel B - MK-8150 4 to 120 mg/Placebo (N=8) | Panel C - MK-8150 5 to 90 mg/Placebo (N=8) | Panel D - MK-8150 50 to 200 mg (N=8) | Panel D - Placebo (N=2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (6) | 0 (0) | 2 (2) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (4) | 3 (5) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration of finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia of lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Pain ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (19) | 7 (37) | 6 (10) | 7 (28) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flushes facial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.